CLINICAL TRIAL: NCT02346396
Title: Non-invasive Analgesic Stimulation of the Motor Cortex at Home
Brief Title: Cortical Stimulation by Direct Current for the Treatment of Chronic Pain : Pilot-study of a Stimulation Device at Home
Acronym: STIMATHOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2014.869; 2014-A01437-40 (Other: ID-RCB)
Record Dates: First submitted 2015-01-07; First posted 2015-01-27 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; neurostimulation; ambulatory use; tDCS
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Efficacy will be assessed in a single-blind trial, with each patient receiving a series of "placebo" stimulations to check the clinical reality of the effects on pain.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with neuropathic chronic pain (Experimental)
  Interventions: Device: tDCS (use at home)

INTERVENTIONS:
Device: tDCS (use at home) — During 4 weeks (every week : 20 minutes / day during 5 days)

SUMMARY:
The purpose of this study is to confirm the analgesic effect of tDCS in neuropathic chronic pain, to estimate the importance and the duration of this effect, and to improve its efficiency by the use at home.

It is established that the repetition of the sessions of cortical stimulation over a week improves their analgesic efficacy. However, this effect does not exceed a few weeks and is much lower than that of the stimulation implanted surgically. Implanted stimulation operates periodically, several times a day, and this "repetition of doses ", akin to the regular taking of a medicine, may explain its longer efficacy for pain relief which, may extend over several years (André-Obadia and al 2014).

No study at this date has estimated the long-term effect of non-invasive stimulation when is also periodically repeated on a daily basis, over several weeks.

ELIGIBILITY:
Inclusion Criteria :

* Patients from 18 to 80 years old, men or women, suffering pharmaco-resistant neuropathic chronic pain for more than one year; NVS > 2 during the week S0) unilateral pharmacoresistant, whose analgesic treatment is stable for at least 1 month.
* Patients whose pharmacoresistance leads their referent doctor to consider non-pharmacological therapeutic alternatives and begin a presurgical assessment.
* Patients having an operational Internet connection. The patient or one person of its circle of acquaintances will have to be able to connect on the Internet and to reach by this way the system of relocated stimulation ("The Cloud").
* Patients having shown pain relief to a single- or whole-week sessions of tDCS are not excluded from potential recruitment for this study.
* Patients having a social security cover.
* Patients having given their written consent.

Exclusion Criteria :

* History
* of addiction to drugs,
* of epilepsy.
* Présence of an intra-cranial ferromagnetic equipment or of an implanted stimulation device (e.g. stimulating, central grey pacemaker, stimulation of the basal ganglia or of the vagus nerve).
* Introduction of a new analgesic treatment for less than a month.
* Lack of a effective contraception for all the duration of the study for the patients old enough to procreate.

(No limitation in the inclusion of male patients old enough to procreate).

* Patient under legal protective measure.
* Pregnant women and nursing mothers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-02-09 (Actual); Primary Completion 2027-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep : numerical rating scale (NRS) from 0 (no sleep) to 10 (very good sleep). | over the week preceding the stimulation (W1), the period of ambulatory stimulation (W2-3-4-5) and the month according to the latter (W6-7-8-9-10)
Fatigue : numerical rating scale (NRS) from 0 (exhausted) to 10 (very well) | over the week preceding the stimulation (W1), the period of ambulatory stimulation (W2-3-4-5) and the month according to the latter (W6-7-8-9-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Neurological Hospital - University Pain Clinic (CETD), Bron, France